CLINICAL TRIAL: NCT01436058
Title: Phase 1 Study of Side Effects of Autologous Mesenchymal Stem Cell Transplantation in Patients With Ankle Joint Osteoarteritis
Brief Title: Side Effects of Autologous Mesenchymal Stem Cell Transplantation in Ankle Joint Osteoartritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-007
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2010-05

CONDITIONS: Osteoarthritis
Keywords: side effect; mesenchymal stem cell; ankle; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell recipient (Experimental): patients with ankle joint osteoarthritis
  Interventions: Biological: mesenchymal stem cell

INTERVENTIONS:
Biological: mesenchymal stem cell — intraarticular injection of mesenchymal stem cell in patients with ankle joint osteoarthritis
  Other Names: stem cell transplantation

SUMMARY:
Ankle osteoarthritis is a joint condition which results from damage and loss of the cartilage in a joint. Treatment options for ankle osteoarthritis are usually aimed at controlling pain and limiting motion that provokes the pain. Nonsurgical treatment approaches are tried first. If unsuccessful, surgical options are considered. Stem cell therapy is one of the therapeutic options that can repair the damaged cartilage. Bone marrow derived mesenchymal stem cells have showed the capacity of bone and cartilage regeneration.

DETAILED DESCRIPTION:
In this clinical study the investigators aim to investigate the safety of intra-articular injection of cultured autologous bone marrow derived mesenchymal stem cells (BM-MSCs) to the ankle joint in patients with severe ankle osteoarthritis. Patients will undergo bone marrow aspiration and will receive cultured BM-MSCs one month later. Patients will be assessed clinically with scoring system (FAO, VAS, WOMAC) preoperatively as well as 2 and 6 months postoperative to measure pain reduction and joint function improvement. Paraclinical studies (X-Ray and MRI) will be performed before and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis diagnosed by MRI
* End stage osteoarthritis candidate for total ankle replacement

Exclusion Criteria:

* Pregnancy or lactating
* Positive tests for HIV, HCV, HBV
* Active neurologic disorder
* End organ damage
* Uncontrolled endocrine disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
safety | 6 months
  Evaluate Safety of intra-articular injection of autologous cultured mesenchymal stem cells in patients with ankle osteoarthritis (time frame : baseline, 2 months, 6 months)by filling the check list of side effects

SECONDARY OUTCOMES:
pain | 6 months
  evaluation the pain reduction in patients with ankle joint osteoarthritis after stem cell transplantation by filling the SF36
physical function | 6 months
  evaluation the ability of patient to standing,walking,climb the steps after stem cell transplantation.
defect | 6 months
  evaluation regeneration of ankle joint by serial MRI after stem cell transplantation based on changing the size of articular defect

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan Cell therapy Center; Mohsen Emadeddin, MD, Principal Investigator — orthopedic scientists
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Emadedin M, Ghorbani Liastani M, Fazeli R, Mohseni F, Moghadasali R, Mardpour S, Hosseini SE, Niknejadi M, Moeininia F, Aghahossein Fanni A, Baghban Eslaminejhad R, Vosough Dizaji A, Labibzadeh N, Mirazimi Bafghi A, Baharvand H, Aghdami N. Long-Term Follow-up of Intra-articular Injection of Autologous Mesenchymal Stem Cells in Patients with Knee, Ankle, or Hip Osteoarthritis. Arch Iran Med. 2015 Jun;18(6):336-44. PMID 26058927
- See also: Related Info — http://www.royaninstitute.org/cmsen/index.php